CLINICAL TRIAL: NCT03331328
Title: MonaLisa Touch Randomized Double-Blind Placebo Controlled Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Michigan Institution of Women's Health PC (Other)
Responsible Party: Principal Investigator, Salil Khandwala, Dr. Salil Khandwala, MD, FACOG, FPMRS, Michigan Institution of Women's Health PC
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1176303
Record Dates: First submitted 2017-08-31; First posted 2017-11-06 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Genitourinary Syndrome of Menopause
Keywords: MonaLisa; Genitourinary syndrome of menopause (GSM)

STUDY DESIGN:
Intervention Model Description: All subjects will be consented for the study prior to the procedure. They will be made aware of the meaning of case control study. Subjects will be randomized to a treatment or a non-treatment group.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Control/sham (Sham Comparator): The CO2 laser will not be activated but the same procedure of moving the probe inside the vagina in a systematic manner including depressing the foot pedal at similar frequency will be performed. The smoke evacuator will also be activated, laser eye glasses and masks worn by the laser team and the subject. However, the laser will remain in the standby mode.
  Interventions: Device: MonaLisa Touch
- Treated (Active Comparator): Active arm subjects will be treated intravaginally with the fractional microablative CO2 laser system (SmartXide 2 V 2 LR, MonaLisa Touch, DEKA, Florence, Italy), using the following setting: dot power 30 watt, dwell time 1000 μs, dot spacing 1000 μm and the smart stack parameter from 1 to 3. For the vulva, the dot power will be reduced to 26 watts, dwell time 800 μs, dot spacing 800 μm and the smart stack parameter of 1.
  Interventions: Device: MonaLisa Touch

INTERVENTIONS:
Device: MonaLisa Touch — MonaLisa Touch is a fractional CO2 laser that has been specially designed with the DEKA pulse to stimulate vaginal tissue. It is delivered in a very precise manner and results in the synthesis of collagen and stratification of the vaginal epithelium with improvement of the vaginal pH and moisturization of the vaginal tissue due to increased blood flow and turgidity of the ground substance from the synthesis of the proteoglycans, hyaluronic acid and collagen.

SUMMARY:
Aim of the study: To assess the efficacy of MonaLisa Touch procedure for the management of genitourinary syndrome of menopause (GSM) in a randomized double-blind placebo controlled study.

DETAILED DESCRIPTION:
Study design: Randomly assigning the intervention can eliminate the influence of unknown or immeasurable confounding variables that may otherwise lead to biased and incorrect estimate of treatment effect. Also, randomization eliminates confounding by baseline variables and blinding eliminates confounding by co-interventions, thus eliminating the possibility that the observed effects of intervention are due to differential use of other treatments. The best comparison is placebo control that allows participants, investigators and study staff to be blinded. The advantage of trial over an observational study is the ability to demonstrate causality.

Background: Genitourinary syndrome of Menopause is a condition of postmenopausal women due to estrogen deprivation which results in progressive worsening of the vaginal and vulvar anatomy with symptoms of vulvar itching or pain during intercourse, vaginal dryness, urinary urgency and frequency and frequent bladder infections. It could ultimately lead to vaginal bleeding, petechial hemorrhages, vaginal narrowing or stenosis and hypertonicity of the pelvic muscles due to anticipation of coital pain. The hypertonicity by itself can cause pelvic pressure or pain.

Thus, GSM is a chronic progressive disease state that if left untreated could have dire vaginal and urogynecological consequences.

MonaLisa Touch is a fractional CO2 laser that has been specially designed with the DEKA pulse to stimulate vaginal tissue. It is delivered in a very precise manner and results in the synthesis of collagen and stratification of the vaginal epithelium with improvement of the vaginal pH and moisturization of the vaginal tissue due to increased blood flow and turgidity of the ground substance from the synthesis of the proteoglycans, hyaluronic acid and collagen.

Initial trials on MonaLisa Touch have shown promising results with significant improvement in vaginal exams and patient satisfaction scores.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal dyspareunia or vaginal dryness rated from moderate to severe
* Desirous of sexual function
* Menopausal women with absence of menstruation for at least 12 months or those who have had bilateral oophorectomy
* Presence of vaginal atrophy symptoms based upon the vaginal health index assessment < 15 and vagina pH >5
* Prolapse stage < III, according to the pelvic organ prolapse quantification (POP-Q) system
* No pelvic reconstructive surgery within 6 months prior to treatment
* Understanding and acceptance of the obligation to return for all scheduled follow-up visits

Exclusion Criteria:

* History of vaginal carcinoma or dysplasia, history of vaginal or pelvic radiation
* Acute or recurrent genital infection (e.g. bacterial; vaginosis, herpes genitalis, candida)
* Any serious disease, or chronic condition such as uncontrolled diabetes, that could interfere with the study compliance
* Reconstructive pelvic surgery within the past 6 months
* Have used vaginal estrogen cream, ring or tablet within 3 months prior to entering the study
* Have used vaginal moisturizers, lubricants or homeopathic preparations within 30 14 days of therapy
* Not willing to stop use of any vaginal lubricants or estrogen of any form including phytoestrogens such as Estroven

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2017-09-13 (Actual); Primary Completion 2019-07-10 (Actual); Study Completion 2019-07-10 (Actual)

PRIMARY OUTCOMES:
Improvement of dyspareunia as rated by a severity score of dyspareunia | 1 year
  Improvement in the most bothersome symptom (MBS) of vulvovaginal atrophy as defined by improvement in dyspareunia. Patients are required to rate the severity of dyspareunia/dryness as none, mild, moderate or severe. The severity score is given a numerical value (none 0, mild 1, moderate 2 and severe 3).

SECONDARY OUTCOMES:
Assess improvement of vaginal dryness as rated by a severity score | 1 year
  Improvement in the most bothersome symptom (MBS) of vulvovaginal atrophy as defined by improvement in vaginal dryness. Patients are required to rate the severity of dyspareunia/dryness as none, mild, moderate or severe. The severity score is given a numerical value (none 0, mild 1, moderate 2 and severe 3).
Assess improvement in irritative bladder symptoms (urgency, frequency, or urination) as rated by a severity score | 1 year
  Improvement in irritative bladder symptoms. Patients are required to rate the severity irritative bladder symptoms of as none, mild, moderate or severe. The severity score is given a numerical value (none 0, mild 1, moderate 2 and severe 3).
Assess improvement in vaginal burning as rated by a severity score | 1 year
  Improvement in the vulvovaginal atrophy symptom of burning as defined by improvement in dyspareunia. Patients are required to rate the severity of dyspareunia/dryness as none, mild, moderate or severe. The severity score is given a numerical value (none 0, mild 1, moderate 2 and severe 3).

CONTACTS AND LOCATIONS:
Locations (1):
- Advanced Urogynecology of Michigan, P.C., Dearborn, Michigan, United States